CLINICAL TRIAL: NCT02415751
Title: The Impact of a Heart Failure Review on Self-Care Knowledge, Adherence and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: CHI Nebraska Heart (Unknown)
Responsible Party: Principal Investigator, Katie Packard, Co-Investigator, Creighton University
Other Study IDs: 742726-1
Record Dates: First submitted 2015-04-07; First posted 2015-04-14 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- self-care education: All patients in the study will receive self-care education
  Interventions: Behavioral: heart failure self-care education

INTERVENTIONS:
Behavioral: heart failure self-care education — It is defined as a naturalistic decision-making process that patients use in the choice of behaviors that maintain physiological stability (symptom monitoring and treatment adherence) and the response to symptoms when they occur (Riegel 2004). This includes following advice regarding medications, sodium and water consumption, alcohol restriction, exercise, preventive behaviors, and monitoring of signs and symptoms.

SUMMARY:
This study is assessing the effects of a new heart failure self-care education program in the Nebraska Heart Institute Heart Improvement Clinic. The new education program will consist of an initial intensive self-care education session with the Principal Investigator or her nurse practitioner. Topics to be discussed include medications, sodium and fluid consumption, alcohol restriction, exercise, preventive behaviors, and monitoring of signs and symptoms. As recommended in the ACCF/AHA guidelines, this education will be repeated on an annual basis as studies have shown that the impact of HF education is not always durable and must be a continual process. This study will assess the impact of this review on their medication knowledge, disease state knowledge, quality of life, disease state progression and clinical outcomes such as ejection fraction and number of hospitalizations.

DETAILED DESCRIPTION:
This is an observational study as all patients in the heart failure clinic, regardless of whether or not they will choose to be in the study, will receive heart failure self-care education from now on.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 19 and older
* Able to speak, read and understand English and able to understand and provide informed consent
* Diagnosis of cardiomyopathy and/or HF, preserved or reduced ejection fraction

Exclusion Criteria:

* Patients not-responsible for self-care.
* Inability to provide written informed consent.
* Co-morbid condition with an expected survival of less than six months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults ages 19 and older with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
number of hospitalizations | 12 months

SECONDARY OUTCOMES:
ejection fraction | 12 months
change in heart failure medication knowledge | 12 months
  Adapted from the Atlanta Heart Failure Knowledge Test V2 (AHFKT-VT) (Miller Reilly C 2009) Grading: 1 point for correct answer, 0 points for incorrect or skipped Total points and divide by 6 for percentage score

CONTACTS AND LOCATIONS:
Overall Officials: Katie Packard, PharmD, Principal Investigator — Creighton University
Locations (2):
- United States (2):
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Creighton University, Omaha, Nebraska